CLINICAL TRIAL: NCT00611559
Title: Immunogenicity and Reactogenicity Study of a New Formulation of GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine Administered as a Booster Dose to 18-23 Months Old Children
Brief Title: Study of a New Formulation of DTPa-HBV-IPV/Hib Vaccine Administered as a Booster Dose to 18-23 Months Old Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110478
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2009-08-10 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2017-05

CONDITIONS: Poliomyelitis; Acellular Pertussis; Tetanus; Diphtheria; Hepatitis B
Keywords: Infanrix hexa; combined vaccine
MeSH Terms: conditions — Poliomyelitis; Tetanus; Diphtheria; Hepatitis B | interventions — PEDIARIX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Infanrix hexa Preservative-Free Formulation Group (Experimental): Subjects received a booster dose of the preservative-free formulation of Infanrix™ hexa
  Interventions: Biological: Infanrix™ hexa
- Infanrix hexa Preservative-Containing Formulation Group (Active Comparator): Subjects received a booster dose of the preservative-containing formulation of Infanrix™ hexa
  Interventions: Biological: Infanrix™ hexa
- Infanrix penta Preservative-Free Formulation Group (Active Comparator): Subjects received a booster dose of the preservative-free formulation of Infanrix™ penta.
  Interventions: Biological: Infanrix™ penta

INTERVENTIONS:
Biological: Infanrix™ penta — Subjects received a booster dose
  Other Names: Pediarix
  Arms: Infanrix penta Preservative-Free Formulation Group
Biological: Infanrix™ hexa — Subjects received a booster dose
  Arms: Infanrix hexa Preservative-Containing Formulation Group; Infanrix hexa Preservative-Free Formulation Group

SUMMARY:
The new formulation administered as a 4th consecutive dose will be compared to the current formulation of the vaccine in this partially double blind study.

The study will be double-blind with respect to the two DTPa-HBV-IPV/Hib groups. The study will be open with respect to the DTPa-HBV-IPV group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects must have completed full three-dose primary vaccination course with DTPa-HBV-IPV/Hib or DTPa-HBV-IPV in the primary study DTPa-HBV-IPV-109 (study NCT00320463).
* A male or female between, and including 18 and 23 months of age at the time of the booster vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the booster dose.
* Participation in another clinical study, between the primary study NCT00320463 and the present booster study, or at any time during the study, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against diphtheria, tetanus, pertussis, poliomyelitis and hepatitis B since the conclusion visit of study NCT00320463.
* Previous booster vaccination against Haemophilus influenzae diseases in the DTPa-HBV-IPV/Hib groups, since the conclusion visit of study NCT00320463.
* History of exposure to diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B and/or Haemophilus influenzae disease since the conclusion visit of study NCT00320463.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Any of the following adverse events having occurred after previous administration of DTP vaccine:
* Hypersensitivity reaction due to the vaccine.
* Encephalopathy defined as an acute, severe central nervous system disorder of unknown etiology occurring within 7 days following previous vaccination and generally consisting of major alterations in consciousness, unresponsiveness, generalized or focal seizures that persist more than a few hours, with failure to recover within 24 hours.
* Any of the following adverse events having occurred after previous administration of DTP vaccine:
* Temperature of >= 40.0 °C (axillary temperature), within 48 hours of vaccination.
* Collapse or shock-like state within 48 hours of vaccination.
* Persistent, inconsolable crying lasting >= 3 hours, occurring within 48 hours of vaccination.
* Convulsions with or without fever, occurring within 3 days of vaccination

Ages: 18 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2008-02-14; Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Russia (3):
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Syktyvkar

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Infanrix Hexa Preservative-free Formulation Group: Subjects received a booster dose of the preservative-free formulation of Infanrix hexa
- Infanrix Hexa Preservative-containing Formulation Group: Subjects received a booster dose of the preservative-containing formulation of Infanrix hexa
- Infanrix Penta Preservative-free Formulation Group: Subjects received a booster dose of the preservative-free formulation of Infanrix penta
Period: Overall Study
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Started | 111 | 115 | 57
Completed | 110 | 114 | 56
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group | Total
Number analyzed (Participants) | 111 | 115 | 57 | 283
Age, Continuous [Mean (Standard Deviation); unit: months] | 21.2 (1.61) | 21.3 (1.57) | 21.2 (1.62) | 21.2 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 46 | 35 | 137
  Male | 55 | 69 | 22 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian/European Heritage | 111 | 115 | 57 | 283

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis B (HB) Antibody Concentrations Above the Cut-off One Month After the Booster Dose
Description: Anti-HB antibodies cut-off value assessed was ≥ 10 milli-international units per milliliter (mIU/mL)
Time Frame: One month after the booster dose
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 91 | 92 | 48
subjects | 88 | 92 | 48

2. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol-phosphate (PRP) Antibodies Concentrations Above the Cut-off One Month After the Booster Dose
Description: Anti-PRP antibodies cut-off value assessed was ≥ 0.15 microgram per milliliter (µg/mL)
Time Frame: One month after the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 76 | 79 | 42
subjects | 74 | 78 | 27

3. Primary Outcome: Number of Subjects With Anti-diphtheria and Anti-tetanus Antibodies Concentration Above the Cut-off One Month After the Booster Dose
Description: Anti-diphtheria and anti-tetanus antibodies cut-off value assessed was ≥ 0.1 international units per milliliter (IU/mL)
Time Frame: One month after the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 77 | 79 | 42
subjects
  Anti-diphtheria | 76 | 76 | 40
  Anti-tetanus | 76 | 78 | 42

4. Primary Outcome: Number of Subjects With Anti-poliovirus Antibodies Concentration Above the Cut-off One Month After the Booster Dose
Description: Anti-poliovirus antibodies cut-off value assessed was ≥ 8 effective dose 50 (ED50)
Time Frame: One month after the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 55 | 52 | 31
subjects
  Anti-poliovirus type 1: number analyzed (Participants) | 55 | 51 | 31
  Anti-poliovirus type 1 | 55 | 51 | 31
  Anti-poliovirus type 2: number analyzed (Participants) | 55 | 51 | 31
  Anti-poliovirus type 2 | 55 | 51 | 30
  Anti-poliovirus type 3 | 55 | 52 | 29

5. Primary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibodies Concentration One Month After the Booster Dose
Description: Concentration of anti-PT, ant-FHA and anti-PRN antibodies given as geometric mean concentration (GMC) in Enzyme-Linked Immuno Sorbent Assay (ELISA) unit per millilitre (EL.U/mL)
Time Frame: One month after the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 89 | 77 | 41
EL.U/mL
  Anti-PT: number analyzed (Participants) | 84 | 70 | 33
  Anti-PT | 65.5 [49.8 to 86.3] | 84.2 [61.5 to 115.4] | 43.9 [22.4 to 85.8]
  Anti-FHA: number analyzed (Participants) | 86 | 69 | 38
  Anti-FHA | 476.6 [369.7 to 614.4] | 428.3 [311.2 to 589.5] | 221.1 [120.3 to 406.6]
  Anti-PRN | 418.1 [303.2 to 576.6] | 384.1 [271.3 to 544.0] | 251.6 [143.9 to 439.7]

6. Secondary Outcome: Number of Subjects With Anti-hepatitis B (HB) Antibody Concentrations Above the Cut-off Before and One Month After the Booster Dose
Description: Anti-HB antibodies cut-off value assessed were ≥ 10 mIU/mL and ≥ 100 mIU/mL
  Number of subjects with cut-off ≥ 10 mIU/mL one month after the booster dose was already presented in the primary outcomes
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 93 | 93 | 48
subjects
  ≥ 10 mIU/mL Pre: number analyzed (Participants) | 93 | 93 | 47
  ≥ 10 mIU/mL Pre | 87 | 86 | 44
  ≥ 100 mIU/mL Pre: number analyzed (Participants) | 93 | 93 | 47
  ≥ 100 mIU/mL Pre | 57 | 57 | 35
  ≥ 100 mIU/mL Post: number analyzed (Participants) | 91 | 92 | 48
  ≥ 100 mIU/mL Post | 85 | 87 | 39

7. Secondary Outcome: Anti-HB Antibodies Concentration
Description: Concentration of anti-HB antibodies given as GMC in mIU/mL
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 93 | 93 | 48
mIU/mL
  Pre: number analyzed (Participants) | 93 | 93 | 47
  Pre | 163.5 [114.3 to 233.7] | 161.2 [111.5 to 232.9] | 196.9 [124.2 to 312.2]
  Post: number analyzed (Participants) | 91 | 92 | 48
  Post | 4668.0 [2861.4 to 7615.3] | 4962.3 [3289.7 to 7485.4] | 3867.8 [1751.4 to 8541.5]

8. Secondary Outcome: Number of Subjects With Anti-PRP Antibodies Concentrations Above the Cut-off Before and One Month After the Booster Dose
Description: Anti-PRP antibodies cut-off value assessed were ≥ 0.15 µg/mL and ≥ 1.0 µg/mL
  Number of subjects with cut-off ≥ 0.15 µg/mL one month after the booster dose was already presented in the primary outcomes
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 76 | 79 | 42
subjects
  ≥ 0.15 µg/mL Pre: number analyzed (Participants) | 75 | 72 | 42
  ≥ 0.15 µg/mL Pre | 55 | 55 | 23
  ≥ 1.0 µg/mL Pre: number analyzed (Participants) | 75 | 72 | 42
  ≥ 1.0 µg/mL Pre | 12 | 14 | 7
  ≥ 1.0 µg/mL Post | 69 | 74 | 9

9. Secondary Outcome: Anti-PRP Antibodies Concentration
Description: Concentration of anti-PRP antibodies given as GMC in µg/mL
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 76 | 79 | 42
µg/mL
  Pre: number analyzed (Participants) | 75 | 72 | 42
  Pre | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.5] | 0.2 [0.1 to 0.4]
  Post | 25.3 [16.0 to 40.0] | 34.7 [22.9 to 52.7] | 0.4 [0.2 to 0.7]

10. Secondary Outcome: Number of Subjects With Anti-diphtheria and Anti-tetanus Antibodies Concentration Above the Cut-off Before the Booster Dose
Description: Anti-diphtheria and anti-tetanus antibodies cut-off value assessed was ≥ 0.1 IU/mL
Time Frame: Before the booster dose administration (at baseline)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 75 | 72 | 42
subjects
  Anti-diphtheria | 45 | 47 | 23
  Anti-tetanus | 69 | 62 | 39

11. Secondary Outcome: Anti-diphtheria and Anti-tetanus Antibodies Concentration
Description: Concentration of anti-diphtheria and anti-tetanus antibodies given as GMC in IU/mL
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 77 | 79 | 42
IU/mL
  Anti-diphtheria Pre: number analyzed (Participants) | 77 | 72 | 42
  Anti-diphtheria Pre | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  Anti-diphtheria Post | 2.7 [1.9 to 3.7] | 3.4 [2.5 to 4.5] | 2.2 [1.4 to 3.5]
  Anti-tetanus Pre: number analyzed (Participants) | 75 | 72 | 42
  Anti-tetanus Pre | 0.5 [0.3 to 0.6] | 0.5 [0.3 to 0.7] | 0.3 [0.2 to 0.4]
  Anti-tetanus Post | 4.9 [3.6 to 6.7] | 6.9 [5.3 to 9.0] | 4.5 [2.8 to 7.4]

12. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibodies Concentration Above the Cut-off Before and One Month After the Booster Dose
Description: Anti-PT, anti-FHA and anti-PRN antibodies cut-off value assessed were ≥ 5 EL.U/mL
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 89 | 84 | 43
subjects
  Anti-PT Pre: number analyzed (Participants) | 83 | 84 | 42
  Anti-PT Pre | 45 | 43 | 26
  Anti-PT Post: number analyzed (Participants) | 84 | 70 | 33
  Anti-PT Post | 79 | 66 | 25
  Anti-FHA Pre: number analyzed (Participants) | 85 | 77 | 42
  Anti-FHA Pre | 77 | 68 | 39
  Anti-FHA Post: number analyzed (Participants) | 83 | 69 | 38
  Anti-FHA Post | 86 | 69 | 37
  Anti-PRN Pre: number analyzed (Participants) | 85 | 84 | 43
  Anti-PRN Pre | 75 | 67 | 35
  Anti-PRN Post: number analyzed (Participants) | 89 | 77 | 41
  Anti-PRN Post | 88 | 77 | 40

13. Secondary Outcome: Anti-PT, Anti-FHA, and Anti-PRN Antibodies Concentration Before the Booster Dose
Description: Concentration of anti-PT, anti-FHA and anti-PRN antibodies given as GMC in EL.U/mL
Time Frame: Before the booster dose administration (at baseline)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 85 | 84 | 43
EL.U/mL
  Anti-PT: number analyzed (Participants) | 83 | 78 | 42
  Anti-PT | 6.6 [5.2 to 8.4] | 6.2 [5.0 to 7.8] | 7.1 [5.3 to 9.4]
  Anti-FHA: number analyzed (Participants) | 85 | 77 | 42
  Anti-FHA | 24.5 [18.4 to 32.6] | 22.1 [16.3 to 30.0] | 23.8 [17.3 to 32.6]
  Anti-PRN | 17.5 [13.4 to 23.0] | 13.7 [10.3 to 18.1] | 15.0 [10.3 to 21.9]

14. Secondary Outcome: Number of Subjects With Anti-poliovirus Antibodies Concentration Above the Cut-off Before the Booster Dose
Description: Anti-poliovirus antibodies cut-off value assessed was ≥ 8 ED50
Time Frame: Before the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 49 | 51 | 27
subjects
  Anti-poliovirus type 1: number analyzed (Participants) | 49 | 50 | 26
  Anti-poliovirus type 1 | 46 | 47 | 24
  Anti-poliovirus type 2: number analyzed (Participants) | 49 | 50 | 27
  Anti-poliovirus type 2 | 46 | 48 | 26
  Anti-poliovirus type 3 | 47 | 48 | 23

15. Secondary Outcome: Anti-poliovirus Antibodies Titer
Description: Concentration of anti-poliovirus antibodies given as geometric mean titers (GMT)
Time Frame: Before (Pre) and one month after (Post) the booster dose
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 55 | 51 | 31
titer
  Anti-poliovirus type 1 Pre: number analyzed (Participants) | 49 | 50 | 26
  Anti-poliovirus type 1 Pre | 106.5 [67.9 to 167.0] | 120.4 [76.9 to 188.4] | 85.9 [47.1 to 156.5]
  Anti-poliovirus type 1 Post | 1237.1 [940.7 to 1626.9] | 1939.8 [1465.1 to 2568.2] | 979.5 [539.4 to 1778.8]
  Anti-poliovirus type 2 Pre: number analyzed (Participants) | 49 | 50 | 27
  Anti-poliovirus type 2 Pre | 144.4 [96.9 to 215.2] | 102.5 [68.2 to 154.2] | 95.3 [56.3 to 161.1]
  Anti-poliovirus type 2 Post | 1412.0 [1096.4 to 1818.5] | 1900.6 [1399.7 to 2580.7] | 916.3 [498.1 to 1685.5]
  Anti-poliovirus type 3 Pre: number analyzed (Participants) | 49 | 51 | 27
  Anti-poliovirus type 3 Pre | 98.7 [68.0 to 143.2] | 68.9 [47.0 to 101.1] | 77.5 [41.9 to 143.4]
  Anti-poliovirus type 3 Post: number analyzed (Participants) | 49 | 51 | 27
  Anti-poliovirus type 3 Post | 1485.9 [1041.4 to 2120.3] | 1828.7 [1303.8 to 2565.1] | 605.6 [264.0 to 1389.1]

16. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include drowsiness, fever, irritability, and loss of appetite
Time Frame: Within the 4-day (Day 0-3) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 111 | 115 | 57
subjects
  Pain | 35 | 36 | 14
  Redness | 54 | 54 | 22
  Swelling | 39 | 45 | 19
  Drowsiness | 21 | 18 | 8
  Fever | 18 | 15 | 6
  Irritability | 21 | 21 | 4
  Loss of appetite | 22 | 14 | 5

17. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within the 31-day (Day 0-30) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 111 | 115 | 57
subjects | 8 | 9 | 2

18. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above
Time Frame: Up to one month after the booster dose administration
Measure: Number; unit: subjects
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
Number analyzed (Participants) | 111 | 115 | 57
subjects | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Infanrix Hexa Preservative-free Formulation Group | Infanrix Hexa Preservative-containing Formulation Group | Infanrix Penta Preservative-free Formulation Group
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/115 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/115 | 0/57
Other Adverse Events (participants affected / at risk) | 59/111 | 62/115 | 26/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Hexa Preservative-free Formulation Group (N=111) | Infanrix Hexa Preservative-containing Formulation Group (N=115) | Infanrix Penta Preservative-free Formulation Group (N=57)
Pain (General disorders) | 35 | 36 | 14
Redness (General disorders) | 54 | 54 | 22
Swelling (General disorders) | 39 | 45 | 19
Drowsiness (General disorders) | 21 | 18 | 8
Fever (General disorders) | 18 | 15 | 6
Irritability (General disorders) | 21 | 21 | 4
Loss of appetite (General disorders) | 22 | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.